CLINICAL TRIAL: NCT02429193
Title: An Open-label Phase 2 Multi-center Study of Enzalutamide and Abiraterone and Biomarkers of Androgen Response and Resistance During Rising PSA: BARRIER-P Trial
Brief Title: Biomarkers of Androgen Response and Resistance In Evolution During a Rising PSA
Acronym: BARRIER-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BARRIER-P
Record Dates: First submitted 2015-03-25; First posted 2015-04-29 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — abiraterone; Prednisone; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone / enzalutamide (Experimental): Abiraterone + prednisone; Enzalutamide
  Interventions: Drug: Abiraterone + prednisone; Drug: Enzalutamide

INTERVENTIONS:
Drug: Abiraterone + prednisone — Abiraterone acetate (1000 mg/day p.o.) + prednisone (5 mg b.i.d., p.o.)
  Other Names: abiraterone acetate; Zytiga; prednisone
Drug: Enzalutamide — Enzalutamide (160 mg/day p.o.)
  Other Names: Xtandi

SUMMARY:
This is an open-label phase 2 multi-center study of abiraterone and enzalutamide in men with castration-resistant prostate cancer. Sixteen patients will be enrolled over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed prostate cancer
* Able to read and understand the consent form, either alone or with the aid of a translator
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nmol/L). If the patient is being treated with luteinizing hormone-releasing hormone (LHRH) agonists (patients who have not undergone orchiectomy), they must remain on continuous androgen suppression therapy throughout the study
* Patients receiving bone-targeted therapies must be on stable doses for at least 4 weeks prior to enrollment
* Historical frozen/paraffin-embedded diagnostic tissue specimens are available for analysis (i.e. radical prostatectomy or biopsy tissue)
* Documented metastatic disease by positive bone scan or metastatic lesions (on CT or MRI) that can be biopsied with an anticipated minimum of 4 cores, as assessed by the local radiologist
* prostate cancer progression at study entry defined as one or more of the following criteria: i. Rising PSA: minimum of two rising PSA levels with an interval of ≥ 1 week between each determination ii. Soft tissue disease progression, as defined by RECIST 1.1 iii. Bone disease progression, as defined by PCWG2 with two or more new lesions on bone scan
* PSA value at screening visit ≥ 2 µg/L (2 ng/mL)
* ECOG performance status 0-2
* Adequate organ and BM function, as defined by the following criteria:

  i. absolute neutrophil count ≥1,500/µL ii. platelets ≥100,000/µL iii. total bilirubin ≤1.5 × institutional upper limit of normal (ULN) iv. AST(SGOT) or ALT(SGPT) ≤2.5 × institutional ULN v. creatinine ≤1.5 × institutional ULN or below
* Serum albumin ≥ 3.0 g/dL
* Serum potassium ≥ 3.5 mmol/L
* Haemoglobin ≥ 10.0 g/dL, independent of transfusion
* Asymptomatic or mildly symptomatic from prostate cancer
* Life expectancy of > 6 months
* Able to swallow study drugs
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 13 weeks after last study drug administration

Exclusion Criteria:

* Patients with known hypersensitivity or allergy to abiraterone acetate, enzalutamide or any of their excipients.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure (NYHA Class 3 or greater), cirrhosis with a Child-Pugh level of B or greater or evidence of cardiac dysfunction, unstable angina pectoris, cardiac arrhythmia, myocardial infarction within 6 months, hypotension (defined by systolic blood pressure < 86 mmHg at Screening visit), hypertension (defined by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at Screening visit), bradycardia (defined by < 50 beats per minute on ECG performed at screening), active peptic ulcer disease, clinically significant gastrointestinal conditions (e.g. Crohns disease, ulcerative colitis), any seizure disorder or psychiatric illness, and social situations that would limit compliance with study requirements
* Active invasive malignancy at any other site excluding squamous cell or basal cell carcinomas of the skin
* Known or suspected brain metastasis or leptomeningeal disease
* Radiotherapy within the past 4 weeks, except for low dose palliative radiation to bone of ≤5 fractions
* Treatment with 5-α reductase inhibitors (finasteride, dutasteride), androgen receptor antagonists (bicalutamide, nilutamide, flutamide), estrogens, cyproterone within 4 weeks of Day 1 visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in expression of androgen receptor abnormalities (e.g. ARV7, AR mutations) following abiraterone/enzalutamide treatment | 18 months
  The change in protein expression of androgen receptor (AR7) splice variant and AR / AR pathway mutations as a mechanism of resistance to abiraterone/enzalutamide is evaluated by measuring the difference in a quantitative immunohistochemical biomarker between assays performed before and after treatment.

SECONDARY OUTCOMES:
Rate of PSA increase | 18 months
Time to PSA progression | 18 months
  PSA progression is defined as a ≥ 25% increase and an absolute increase of ≥ 2 µg/L (2 ng/mL) above the nadir.

OTHER OUTCOMES:
Number of participants with adverse events from the administration of abiraterone, enzalutamide, and prednisone to men with early stage prostate cancer. | 18 months
  The number of participants experiencing adverse events will be evaluated to determine the safety of abiraterone, enzalutamide, and prednisone treatment in men with early stage prostate cancer, .

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, MD,MBBS,PhD,FRACP, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - British Columbia Cancer Agency, Vancouver Cancer Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario